CLINICAL TRIAL: NCT01664273
Title: Gene Electrotransfer to Muscle With Plasmid AMEP in Patients With Disseminated Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Production of the IMP (plasmid AMEP) has been terminated by the supplier (BioAlliance Pharma)
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AA 1201
Record Dates: First submitted 2012-07-16; First posted 2012-08-14 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Metastatic Malignant Neoplasm
Keywords: electroporation; gen electrotransfer; muscle; plasmid AMEP
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Plasmid AMEP — Cohorts of 3 patients will received increasing doses of plasmid AMEP:
  50 μg, 100 μg, 250 μg and 500 μg. Starting dose will be the lowest dose.
  Injection volume will remain constant at 200 μL.
  Once-only treatment and intra-individual dose escalation will therefore not occur.

SUMMARY:
Gene transfer by electroporation (gene electrotransfer) uses short electric pulses to transiently permeabilise the cell membrane enabling passage of plasmid DNA into the cell cytosol. It is an efficient non-viral method for gene delivery to various tissues. In this phase I dose-escalating study, patients will be treated with intramuscular gene electrotransfer of plasmid AMEP. Plasmid AMEP encodes protein AMEP which bind to α5β1 og αvβ3 integrins. Primary end point of the trial is safety and secondary end points are efficacy, pharmacokinetics and evaluation of potential discomfort associated with the treatment procedure using VAS (Visual Analogue Scale).

DETAILED DESCRIPTION:
Cohorts of 3 patients will be treated with increasing doses of plasmid AMEP. Up to 12 patients will be treated.

Treatment procedure: Local anesthetic is applied to m. quadriceps femoris (thigh muscle) and the skin. An incision of the skin is performed followed by dissection until the muscle is exposed. The surgical procedure is performed by plastic surgeons.

Plasmid AMEP is injected intramuscularly and immediately followed by application of electric pulses via a needle electrode inserted into the muscle. A combination of one high voltage pulse (700V/cm, 100 µs) followed by one low voltage pulse (80 V/cm, 400 ms) will be applied. The wound is sutured and a dressing is applied. Treatment procedure is estimated to 30 minutes.

All patients are hospitalized for 24 hours after treatment for the purpose of evaluation of vital signs, physical examination, AE and SAE recording and pharmacokinetics sampling (blood and urine).

Blood biochemistry including LDH and CK is taken 24 hours post treatment. ECG will be taken before and after treatment. Patients score discomfort or pain from treated area using VAS.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Performance status < 1 (ECOG).
* Histologically confirmed malignant tumor (solid tumor) of any histology,
* Metastatic disease. Patients with asymptomatic brain metastases are eligible.
* Patient should have been offered standard treatment. Patient is eligible if no standard treatment is available or if the patient does not wish to receive standard treatment.
* Life expectancy ≥ 3 months.
* Measurable disease defined as at least one measurable lesion according to RECIST 1.1
* Patient should have adequate organ function:
* Adequate bone marrow function: Neutrophil count ≥ 1.0 x 109/l (≤ grade 2 CTCAE 4.0); Platelet count ≥ 75 x 109/l (< grade 2 CTCAE 4.0); Hemoglobin ≥ 6,0 mmol/l.
* Liver: ALAT or ASAT < 3 ULN (< grade 2 CTCAE 4.0); Bilirubin ≤ 1,5 ULN (< grade 2 CTCAE 4.0); APTT within normal range; INR ≤ 1,2 (< grade 1 CTCAE 4.0)
* Kidney: Plasma creatinin ≤ 1.5 ULN (< grade 2 CTCAE 4.0)
* At least 4 weeks since any anti-cancer treatment.
* Men and women of reproductive age must use effective contraception during the study and at least 6 months after administration of plasmid AMEP.
* Patient should be able to understand the participant information and able to comply with protocol requirements and scheduled visits.
* Signed informed consent.

Exclusion Criteria:

* Allergy to the anaesthetic used.
* Clinical signs of active infection.
* Implanted pacemaker, defibrillator or any other implanted electronic device.
* Participation in other clinical trials involving experimental drugs or participation in a clinical trial within 4 weeks before initiation of study treatment.
* AMI (acute myocardial infarction), stroke or acute ischemic event within the last 6 months.
* Severe atherosclerosis, significant cardiovascular disease (NYHA III or IV) or significant arrhythmias.
* Systolic blood pressure above 180 mm Hg and/or diastolic blood pressure above 110 mm Hg. If BP >180/110 mm Hg medical correction is allowed and the patient can be included when BP < 180/110 mm Hg.
* Pregnancy and lactation.
* Clinically significant coagulopathy.
* Treatment with anticoagulant drugs.
* Other disorders which the investigator finds incompatible with participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-07; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Safety of the trial treatment | From treatment to last follow up, planned 8 weeks.
  Safety is evaluated by registration of adverse events (Adverse Events and Serious Adverse Events) using the CTCAE criteria version 4.0. Patients are seen in the out patient clinic once a week during the first month after treatment (at day 8, day 15, day 22, day 29) and 8 weeks after treatment. If no progression of the disease at 8 weeks, patients are seen at 12 weeks and then every three months until disease progression or death.

SECONDARY OUTCOMES:
Efficacy of the trial treatment | PET/CT scan 4 weeks, 8 weeks and 12 weeks after trial treatment.
  PET/CT scan will be evaluated using RECIST 1.1 (CT) and PERCIST (PET)
Pharmacokinetics | Pre-dose, 2, 6 and 24 hours after dose, day 8, 15, 22, 29 and 8 weeks after treatment.
  Measurements of plasma and urine plasmid AMEP concentrations. Measurements of plasma and urine protein AMEP concentrations
Discomfort associated with the treatment procedure | Scoring 'immediately after treatment', '30 min after treatment' '6 hours after treatment' and 'pain in the past 24 hours', and day 8.
  The patient completes VAS (Visual Analogue Scale) scores pain related to the treatment area at abovementioned time points.
Safety | Day after treatment and 14 days after treatment
  MR scan of treated region (thigh muscle) in order to assess potential intramuscular edema or hematoma

CONTACTS AND LOCATIONS:
Overall Officials: Julie Gehl, MD DMSci, Principal Investigator — Department of Oncology, Copenhagen University Hospital Herlev
Locations (1):
- Depart. of Oncology, Copenhagen Universtiy Hospital Herlev, Herlev, Denmark